CLINICAL TRIAL: NCT01205659
Title: Allergy and Asthma in Children Who Were Fed Supplemented Infant Formula (3-7 Years of Age)
Brief Title: Allergy and Ashthma in Children Who Were Fed Supplemented Infant Formula
Status: Completed | Type: Observational
Sponsor: Mead Johnson Nutrition (Industry)
Responsible Party: Eileen Birch, The Retina Foundation of the Southwest
Other Study IDs: 8611
Record Dates: First submitted 2010-09-17; First posted 2010-09-20 (Estimated); Last update posted 2010-09-20 (Estimated); Status verified 2010-09

CONDITIONS: Allergy and Asthma
MeSH Terms: conditions — Hypersensitivity; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Allergy and Asthma study of children (3 - 7 Years of age) who participated in randomized trials of supplemented infant formula during infancy conducted by The Retina Foundation of the Southwest .

ELIGIBILITY:
Inclusion Criteria:

* Children who participated in randomized trials of supplemented infant formula conducted by The Retina Foundation of the Southwest during infancy

Exclusion Criteria:

-

Ages: 3 Years to 7 Years | Sex: All
Age Groups: Child
Study Population: Children who participated in randomizaed trials of supplemented infant formula conducted by The Retina Foundation of the Southwest during infancy
Sampling Method: Probability Sample
Dates: Start 2008-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of asthma and allergy related diagnosis in medical records for ages 3 - 7 years

SECONDARY OUTCOMES:
Prevalence of Serious Adverse Events in medical records
Long-term growth

CONTACTS AND LOCATIONS:
Locations (1):
- The Retina Foundation of The Southwest, Dallas, Texas, United States